CLINICAL TRIAL: NCT01086384
Title: A Long-Term, Randomized, Double-Blind, Parallel Group Study of Fluticasone Furoate/GW642444 Inhalation Powder Once-Daily and Fluticasone Furoate Inhalation Powder Once-Daily in Subjects With Asthma
Brief Title: Asthma Exacerbation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 106837
Record Dates: First submitted 2010-03-11; First posted 2010-03-15 (Estimated); Results first posted 2013-09-11 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluticasone furoate/GW642444 (Experimental)
  Interventions: Drug: Fluticasone Furoate/GW642444
- fluticasone furoate (Experimental)
  Interventions: Drug: Fluticasone furoate

INTERVENTIONS:
Drug: Fluticasone Furoate/GW642444 — Combination inhaled corticosteroid and long-acting beta2-agonist
  Arms: Fluticasone furoate/GW642444
Drug: Fluticasone furoate — Inhaled corticosteroid
  Arms: fluticasone furoate

SUMMARY:
This study will establish the safety as well as demonstrate benefit of the addition of a LABA to an ICS by utilizing an endpoint (time to first severe asthma exacerbation) that informs on both safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma
* Reversibility FEV1 of twelve percent or greater and two hundred milliliters and greater approximately ten to forty minutes following two to four inhalations of albuterol
* FEV1 of fifty to ninety percent of predicted
* Currently using inhaled corticosteroid therapy
* History of one or more asthma exacerbations requiring treatment with oral/systemic corticosteroids or emergency department visit or in-patient hospitalization in previous year

Exclusion Criteria:

* History of life threatening asthma in previous 5 years (requiring intubation, and/or associated with hypercapnia, hypoxic seizure or respiratory arrest
* Respiratory infection or oral candidiasis
* - Uncontrolled disease or clinical abnormality
* Allergies
* Taking another investigational medication or prohibited medication

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2020 (Actual)
Dates: Start 2010-02-22; Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (151):
- United States (61):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Oxford, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Bell Gardens, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Napa, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Cocoa, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Valrico, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Albany, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Lawrenceville, Georgia
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, River Forest, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Hazard, Kentucky
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Rockville Centre, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Sylvania, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Collegeville, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, South Burlington, Vermont
  - GSK Investigational Site, Bellingham, Washington
  - GSK Investigational Site, La Crosse, Wisconsin
- Argentina (6):
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Paraná, Entre Ríos Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (6):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Hornsby, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Toorak Gardens, South Australia
  - GSK Investigational Site, Clayton, Victoria
- Germany (24):
  - GSK Investigational Site, Deggingen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Aschaffenburg, Bavaria
  - GSK Investigational Site, Großheirath, Bavaria
  - GSK Investigational Site, Vilshofen, Bavaria
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Rüdersdorf, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Marburg, Hesse
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Dortmund, North Rhine-Westphalia
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Gelsenkirchen, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Solingen, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Rhaunen, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Erfurt, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Japan (7):
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- Mexico (5):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Monterrey NL, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
  - GSK Investigational Site, Mexico City
- Philippines (4):
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Lipa City
  - GSK Investigational Site, Marilao, Bulacan
  - GSK Investigational Site, Quezon City
- Poland (12):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Koszalin
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Rzeszów
  - GSK Investigational Site, Wołomin
  - GSK Investigational Site, Wroclaw
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Sibiu
- Russia (14):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Penza
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Volgodonsk
  - GSK Investigational Site, Voronezh
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Yalta
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Gross AS, Goldfrad C, Hozawa S, James MH, Clifton CS, Sugiyama Y, Jacques L. Ethnic sensitivity assessment of fluticasone furoate/vilanterol in East Asian asthma patients from randomized double-blind multicentre Phase IIb/III trials. BMC Pulm Med. 2015 Dec 24;15:165. doi: 10.1186/s12890-015-0159-z. PMID 26704701
- [Derived] Bateman ED, O'Byrne PM, Busse WW, Lotvall J, Bleecker ER, Andersen L, Jacques L, Frith L, Lim J, Woodcock A. Once-daily fluticasone furoate (FF)/vilanterol reduces risk of severe exacerbations in asthma versus FF alone. Thorax. 2014 Apr;69(4):312-9. doi: 10.1136/thoraxjnl-2013-203600. Epub 2013 Nov 19. PMID 24253831
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106837 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (par.) who met all entry criteria at Screening entered a 2-week Run-in Period for completion of Baseline safety evaluations and to obtain Baseline measures of asthma status. Participants who met continuation criteria at the end of the Run-in Period were randomized to receive study treatment.
Groups:
- FP 250 µg/ICS: Japanese participants using fluticasone propionate (FP)/salmeterol 250/50 micrograms (µg) twice daily received open-label FP 250 µg to ensure they continued their inhaled corticosteroid (ICS) therapy at a fixed dose during the 2-week Run-in Period. All other participants continued to use their current ICS therapy at a fixed dose during the 2-week Run-in Period. Short-acting beta2-agonist inhalation aerosol (albuterol/salbutamol) was provided to be used as needed for symptomatic relief of asthma symptoms during the Run-in Period.
- FF 100 µg: Participants received fluticasone furoate (FF) 100 microgram (µg) inhalation powder via a dry powder inhaler (DPI) once daily in the evening. Short-acting beta2-agonist inhalation aerosol (albuterol/salbutamol) was provided to be used as needed for symptomatic relief of asthma symptoms during the Treatment Period.
- FF/VI 100/25 µg: Participants received FF/vilanterol (VI) 100/25 µg inhalation powder via a DPI once daily in the evening. Short-acting beta2-agonist inhalation aerosol (albuterol/salbutamol) was provided to be used as needed for symptomatic relief of asthma symptoms during the Treatment Period.
Period: 2-week Run-in Period
Arm/Group | FP 250 µg/ICS | FF 100 µg | FF/VI 100/25 µg
Started | 2183 | 0 | 0
Completed | 2020 | 0 | 0
Not Completed | 163 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Physician Decision | 6 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 0 | 0
Not completed — Study Closed/Terminated | 42 | 0 | 0
Not completed — Continuation Criteria Not Met | 92 | 0 | 0
Not completed — Randomized in Error | 1 | 0 | 0
Period: Treatment Period
Arm/Group | FP 250 µg/ICS | FF 100 µg | FF/VI 100/25 µg
Started | 0 | 1011 | 1009
Completed | 0 | 863 | 885
Not Completed | 0 | 148 | 124
Not completed — Withdrawal by Subject | 0 | 53 | 55
Not completed — Protocol Violation | 0 | 26 | 17
Not completed — Lack of Efficacy | 0 | 22 | 13
Not completed — Adverse Event | 0 | 19 | 15
Not completed — Lost to Follow-up | 0 | 11 | 9
Not completed — Physician Decision | 0 | 9 | 6
Not completed — Study Closed/Terminated | 0 | 7 | 8
Not completed — Protocol-Defined Stopping Criteria | 0 | 0 | 1
Not completed — Received Treatment in Error | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF 100 µg | FF/VI 100/25 µg | Total
Number analyzed (Participants) | 1010 | 1009 | 2019
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristic data were collected in members of the Intent-to-Treat Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
  Years | 42.3 (16.82) | 41.1 (17.10) | 41.7 (16.96)
Sex: Female, Male [Count of Participants; unit: Participants] — Baseline characteristic data were collected in members of the Intent-to-Treat Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
  Participants
    Female | 689 | 661 | 1350
    Male | 321 | 348 | 669
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristic data were collected in members of the Intent-to-Treat Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
  participants
    African American/African Heritage | 47 | 40 | 87
    American Indian or Alaska Native | 4 | 9 | 13
    Asian - Central/South Asian Heritage | 0 | 2 | 2
    Asian - East Asian Heritage | 1 | 0 | 1
    Asian - Japanese Heritage | 30 | 32 | 62
    Asian - South East Asian Heritage | 79 | 78 | 157
    Native Hawaiian or other Pacific Islander | 2 | 0 | 2
    White - Arabic/North African Heritage | 5 | 2 | 7
    White - White/Caucasian/European Heritage | 738 | 738 | 1476
    Mixed Race | 104 | 108 | 212

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 1 or More Severe Asthma Exacerbations
Description: Asthma is a medical condition that causes narrowing of the small airways in the lungs. A severe asthma exacerbation is defined as a deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. Only events deemed by the adjudication committee to be severe asthma exacerbations were used in the analysis of severe asthma exacerbations. The time to the first severe asthma exacerbation was analyzed using a Cox proportional hazards regression model, adjusting for Baseline disease severity (Baseline forced expiratory volume in one second [FEV1, maximum amount of air forcefully exhaled in one second]), sex, age, and region.
Time Frame: Baseline to Follow-up (up to 76 weeks of treatment)
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment who received at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | FF 100 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 1010 | 1009
participants | 186 | 154
Statistical Analysis 1: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; Regression Cox = 0.795, 95% CI 2-sided [0.642 to 0.985] — The estimated values is the Hazard ratio obtained from the Cox regression analysis for FF/VI 100/25 µg versus FF 100 µg, adjusted for an interim analysis
Statistical Analysis 2: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.036, Regression, Cox — P-value for the Hazard ratio obtained from the Cox regression analysis for FF/VI 100/25 µg versus FF 100 µg, adjusted for an interim analysis; Hazard Ratio (HR) = 15.9, 95% CI 2-sided [13.5 to 18.2] — The estimated value represents the adjusted probability of 1 or more severe asthma exacerbations by Week 52 for FF 100 µg. Cox Proportional Hazards Model estimate at mean Baseline FEV1, age, and proportional coefficients for sex and region
Statistical Analysis 3: Comparison: FF 100 µg vs FF/VI 100/25 µg; Test type: Superiority or Other; p = 0.036, Regression, Cox — [p-value comment as in outcome 1, analysis 2]; Cox Proportional Hazard = 12.8, 95% CI 2-sided [10.7 to 14.9] — The estimated value represents the adjusted probability of 1 or more severe asthma exacerbations by Week 52 for FF/VI 100/25 µg. Cox Proportional Hazards Model estimate at mean Baseline FEV1, age, and proportional coefficients for sex and region

2. Secondary Outcome: Number of Severe Asthma Exacerbations
Description: A severe asthma exacerbation is defined as a deterioration of asthma requiring the use of systemic corticosteroids (tablets, suspension, or injection) for at least 3 days or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids. A participant may have had one or more exacerbations.
Time Frame: Baseline to Follow-up (up to 76 weeks of treatment)
Population: ITT Population
Measure: Number; unit: Severe asthma exacerbations
Arm/Group | FF 100 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 1010 | 1009
Severe asthma exacerbations | 271 | 200

3. Secondary Outcome: Change From Baseline in Evening Pre-dose Trough FEV1 at Week 36
Description: Evening pre-dose trough (lowest value) forced expiratory volume in one second (FEV1) was measured using spirometry equipment that met or exceeded the minimal performance recommendations of the American Thoracic Society. FEV1 is a measure of the maximum amount of air forcefully exhaled in one second. Change from Baseline in evening pre-dose FEV1 was analyzed using an Analysis of Covariance (ANCOVA) model with effects due to Baseline FEV1, sex, age, region, and treatment. Change from Baseline was calculated as the Week 36 value minus the Baseline value.
Time Frame: Baseline and Week 36
Population: ITT Population. Only those participants available at the indicated time point (Week 36) were analyzed.
Measure: Least Squares Mean (Standard Deviation); unit: Liters
Arm/Group | FF 100 µg | FF/VI 100/25 µg
Number analyzed (Participants) | 902 | 926
Liters | 0.265 (0.014) | 0.348 (0.014)

ADVERSE EVENTS:
Description: Serious adverse events (SAEs) and non-serious AEs are reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of study medication.
Arm/Group | FF 100 µg | FF/VI 100/25 µg
Serious Adverse Events (participants affected / at risk) | 29/1010 | 41/1009
Other Adverse Events (participants affected / at risk) | 479/1010 | 467/1009
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg (N=1010) | FF/VI 100/25 µg (N=1009)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 4
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Meningitis viral (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Tachyarrthmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Diabetic microangiopathy (Vascular disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Fear (Psychiatric disorders) | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg (N=1010) | FF/VI 100/25 µg (N=1009)
Nasopharyngitis (Infections and infestations) | 131 | 155
Upper respiratory tract infection (Infections and infestations) | 93 | 73
Bronchitis (Infections and infestations) | 74 | 59
Influenza (Infections and infestations) | 38 | 50
Sinusitus (Infections and infestations) | 38 | 42
Pharyngitis (Infections and infestations) | 41 | 29
Headache (Nervous system disorders) | 179 | 188
Cough (Respiratory, thoracic and mediastinal disorders) | 64 | 55
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 55 | 41
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 26 | 39
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26 | 33
Back pain (Musculoskeletal and connective tissue disorders) | 40 | 41
Abdominal pain upper (Gastrointestinal disorders) | 23 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.